CLINICAL TRIAL: NCT01584804
Title: Randomised, Double-blinded, Placebo-Controlled Study of Therapeutic Effect of Su-Huang Antitussive Capsule on Cough Variant Asthma(CVA)
Brief Title: Effects of Su-Huang Antitussive Capsule on Cough Variant Asthma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Kefang Lai, professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003L03253
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Asthma
Keywords: Su Huang antitussive capsule; Cough variant asthma; Placebo
MeSH Terms: conditions — Asthma; Cough-Variant Asthma | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monotherapy (Active Comparator): Monotherapy with Su-Huang antitussive capsule
  Interventions: Drug: Su-Huang antitussive capsule
- Sugar pill (Placebo Comparator): Monotherapy with placebo
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Su-Huang antitussive capsule — Su-Huang antitussive capsule (0.45g) 3 capsules Tid for 2 weeks (swallowed by warm water at 0.5-1h after each meal)
  Arms: Monotherapy
Drug: Sugar pill — Sugar pill 3 capsules Tid for 2 weeks (swallowed by warm water at 0.5-1h after each meal)
  Arms: Sugar pill

SUMMARY:
This study aims to observe the therapeutic effect of Su-Huang antitussive capsule on cough variant asthma.

The investigators hypothesize:

Cough score and cough reflex sensitivity will be improved after treatment with Su-Huang antitussive capsule.

DETAILED DESCRIPTION:
Study groups:

60 patients diagnosed with CVA will be randomised into two groups as follows:

Group 1:Su-Huang antitussive capsule The patients with cough variant asthma received Su-Huang antitussive capsule (0.45g) 3 capsules Tid for 2 weeks (swallowed by warm water at 0.5-1h after each meal).

Group 2: placebo The patients with cough variant asthma received placebo 3 capsules Tid for 2 weeks (swallowed by warm water at 0.5-1h after each meal).

The study will be divided into following phases:

1. First Visit (Visit s, day -14):

   A full medical history and physical examination to be undertaken to determine whether patients meet the inclusion/exclusion criteria.

   After the informed consent has been signed, the following samples are obtained from all patients: blood samples for routine clinical laboratory tests (haematology, biochemistry and electrocardiogram, chest x-ray). A urine pregnancy test will be performed in women of childbearing potential.

   Spirometry and methacholine bronchial provocation test were performed to determined the presence of bronchial non-specific hyper-responsiveness.
2. Screening Period (day -14 to day 0, 14 Days) Patients can take medications other than corticosteroid , β2 agonist, inhaled sodium cromoglycate.
3. Second Visit (Visit 1, Week 0):

   Patients are given the Diary Card.

   A physical examination were to be performed. All laboratory tests results are obtained to determine whether patients meet the inclusion/exclusion criteria. Concurrent medication were recorded.

   Capsaicin challenge test and FENO were performed and hypertonic saline induced sputum samples for cell differential were taken from enrolled patients.

   Enrolled patients were randomized into different groups, and the study medication were dispensed.
4. During Treatment 1(Week 0 to Week 1, 7 days):

   Patients were to take study medication for 14 days and completed Diary Card for 7 days from Week 0 to Week 1.
5. Third Visit (Visit 2, Week 1):

   A physical examination were to be performed. The Diary Card were collected and reviewed. Adverse events, secondary complications, concurrent medication will be recorded.

   The Diary Card were collected, reviewed and assessed whether treatment is efficient for cough symptom (symptom score improved 1 at least).
6. During Treatment 2 (Week 1 to Week 2, 7 days):

Patients were to take study medication for 14 days and completed Diary Card for 7 days from Week 1 to Week 2.

Spirometry and bronchial provocation test by methacholine inhalation,electro-cardiogram,capsaicin challenge test and FENO were performed and hypertonic saline induced sputum samples for cell differential were taken from enrolled patients.

Blood samples for routine clinical laboratory tests (haematology and biochemistry) were obtained, if a clinically significant laboratory abnormal result was noted at the visit 2, AE and a follow-up visit would be considered.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have a history of cough as sole or main symptom lasting more than 8 weeks, often irritating cough more cough at night.
2. Patients who were diagnosed with positive result in bronchial provocation test by methacholine inhalation challenge.
3. There is evidence that bronchodilator treatment* is efficient for cough symptom (symptom score improved 1 at least).
4. Patients whose chest x-ray outcome was normal or without any active focus.
5. Patients who was aged from 18 years old (≥ 18 years old ) to 65 years old (≤ 75 years old).

Exclusion Criteria:

1. Patients demonstrate FEV1/FVC <70% in lung function test. FEV1 stands for forced expiratory volume in 1 second, FVC stands for forced vital capacity.
2. Patients who is a smoker or ex-smoker and has smoked within the previous year or has a cumulative smoking history >10 pack-years or equivalence.
3. Patients with concomitance of GERC (gastroesophageal reflux-related chronic cough), chronic bronchitis , bronchiectasis, bronchial tuberculosis, ACEI induced cough, bronchogenic carcinoma, psychologic cough, pulmonary fibrosis, bronchus foreign body, microlithiasis, tracheobroncheopathia osteochondroplastica, mediastinal tumor, left ventricular dysfunction.
4. Female subjects who are pregnant, breast-feeding or risk of becoming pregnant during the study.
5. Subjects who are known or suspected to be hypersensitive to any component of the study medication or relief medications.
6. Subjects who have received any therapy in the previous seven days, e.g. long-acting β2 agonist, theophylline sustained release.
7. Subjects who have received oral/ inhaled/systematic corticosteroid in the previous 4 weeks.
8. Subjects who are diagnosed with past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, endocrine disease or pulmonary disease. e.g.nasal-sinus infection, lower respiratory tract infection, chronic bronchitis, emphysema, bronchiectasis, cystic fibrosis or bronchopulmonary dysplasia.
9. Subjects who demonstrate significant abnormality on biochemistry, hematology, ECG.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-05 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Day-time and night-time cough symptom total-score changes from baseline to visit 3 | 2 weeks

SECONDARY OUTCOMES:
Cough reflex sensitivity changes in 2 groups at baseline and visit 3. Cell differential changes in hypertonic saline induced sputum in 2 groups at baseline and visit3. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mengfeng Li, MD, Study Chair — Sun Yat-sen University
Locations (1):
- Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong, China